CLINICAL TRIAL: NCT05671822
Title: A Phase Ib/II Study of SHR-A1811 Combinations in Patients With Advanced/Metastatic HER2 Expression Gastric /Gastroesophageal Junction Adenocarcinoma
Brief Title: Ph1b/2 Study of the Safety and Efficacy of SHR-A1811 Combinations in Advanced HER2 Expression Gastric Cancer
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Suzhou Suncadia Biopharmaceuticals Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: SHR-A1811-Ib/II-205
Record Dates: First submitted 2023-01-03; First posted 2023-01-05 (Actual); Last update posted 2026-02-12 (Actual); Status verified 2025-04

CONDITIONS: HER2 Expression Gastric Cancer/Gastroesophageal Junction Adenocarcinoma
MeSH Terms: interventions — SHR-1701; Capecitabine; Fluorouracil

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (12):
- Arm 1A: SHR-A1811 and SHR-1701 (Experimental)
  Interventions: Drug: SHR-A1811 and SHR-1701
- Arm 1B: SHR-A1811 and capecitabine (Experimental)
  Interventions: Drug: SHR-A1811 and capecitabine
- Arm 1C: SHR-A181, SHR-1701, and capecitabine (Experimental)
  Interventions: Drug: SHR-A181, SHR-1701, and capecitabine
- Arm 1D: SHR-A1811, SHR-1316, and capecitabine (Experimental)
  Interventions: Drug: SHR-A1811, SHR-1316, and capecitabine
- Arm 1F: SHR-A1811, SHR-1316, capecitabine,and oxaliplatin (Experimental)
  Interventions: Drug: SHR-A1811, SHR-1316, capecitabine,and oxaliplatin
- Arm 1G: SHR-A1811, SHR-1316, and 5-FU (Experimental)
  Interventions: Drug: SHR-A1811, SHR-1316, and 5-FU
- Arm 2A: SHR-A1811, SHR-1316, and capecitabine (Experimental)
  Interventions: Drug: SHR-A1811, SHR-1316, and capecitabine
- Arm 2B: SHR-1316 and SHR-A181 (Experimental)
  Interventions: Drug: SHR-1316 and SHR-A1811
- Arm 2C: SHR-A1811 and capecitabine (Experimental)
  Interventions: Drug: SHR-A1811 and capecitabine
- Arm 2D: SHR-A1811, SHR-1316, and 5-FU (Experimental)
  Interventions: Drug: SHR-A1811, SHR-1316, and 5-FU
- Arm 2E: SHR-A1811and 5-FU (Experimental)
  Interventions: Drug: SHR-A1811and 5-FU
- Arm 2F: SHR-A1811, SHR-1316, capecitabine,and oxaliplatin (Experimental)
  Interventions: Drug: SHR-A1811, SHR-1316, capecitabine,and oxaliplatin

INTERVENTIONS:
Drug: SHR-A1811 and SHR-1701 — (Arm 1A) Drug: SHR-A1811, administered as an IV infusion Drug: SHR-1701, administered as an IV infusion;
  Arms: Arm 1A: SHR-A1811 and SHR-1701
Drug: SHR-A1811 and capecitabine — (Arm 1B) Drug: SHR-A1811, administered as an IV infusion Drug：capecitabine, administered orally；
  Arms: Arm 1B: SHR-A1811 and capecitabine
Drug: SHR-A181, SHR-1701, and capecitabine — (Arm 1C) Drug: SHR-A1811, administered as an IV infusion Drug: SHR-1701, administered as an IV infusion Drug：capecitabine, administered orally；
  Arms: Arm 1C: SHR-A181, SHR-1701, and capecitabine
Drug: SHR-A1811, SHR-1316, and capecitabine — (Arm 1D) Drug: SHR-A1811, administered as an IV infusion Drug: SHR-1316, administered as an IV infusion Drug：capecitabine, administered orally；
  Arms: Arm 1D: SHR-A1811, SHR-1316, and capecitabine
Drug: SHR-A1811, SHR-1316, capecitabine,and oxaliplatin — (Arm 1F) Drug: SHR-A1811, administered as an IV infusion Drug: SHR-1316, administered as an IV infusion Drug：capecitabine, administered orally； Drug：oxaliplatin，administered as an IV infusion
  Arms: Arm 1F: SHR-A1811, SHR-1316, capecitabine,and oxaliplatin
Drug: SHR-A1811, SHR-1316, and 5-FU — (Arm 1G) Drug: SHR-A1811, administered as an IV infusion Drug: SHR-1316, administered as an IV infusion Drug：5-FU，administered as an IV infusion
  Arms: Arm 1G: SHR-A1811, SHR-1316, and 5-FU
Drug: SHR-A1811, SHR-1316, and capecitabine — (Arm 2A) Drug: SHR-A1811, administered as an IV infusion Drug: SHR-1316 administered as an IV infusion; Drug：capecitabine, administered orally；
  Arms: Arm 2A: SHR-A1811, SHR-1316, and capecitabine
Drug: SHR-1316 and SHR-A1811 — (Arm 2B) Drug: SHR-A1811, administered as an IV infusion Drug: SHR-1316, administered as an IV infusion
  Arms: Arm 2B: SHR-1316 and SHR-A181
Drug: SHR-A1811 and capecitabine — (Arm 2C) Drug: SHR-A1811, administered as an IV infusion Drug：capecitabine, administered orally；
  Arms: Arm 2C: SHR-A1811 and capecitabine
Drug: SHR-A1811, SHR-1316, and 5-FU — (Arm 2D) Drug: SHR-A1811, administered as an IV infusion Drug: SHR-1316, administered as an IV infusion Drug：5-FU，administered as an IV infusion
  Arms: Arm 2D: SHR-A1811, SHR-1316, and 5-FU
Drug: SHR-A1811and 5-FU — (Arm 2E) Drug: SHR-A1811, administered as an IV infusion Drug：5-FU，administered as an IV infusion
  Arms: Arm 2E: SHR-A1811and 5-FU
Drug: SHR-A1811, SHR-1316, capecitabine,and oxaliplatin — (Arm 2F) Drug: SHR-A1811,administered as an IV infusion Drug: SHR-1316, administered as an IV infusion Drug：capecitabine, administered orally； Drug：oxaliplatin，administered as an IV infusion
  Arms: Arm 2F: SHR-A1811, SHR-1316, capecitabine,and oxaliplatin

SUMMARY:
This is an open,multicentre phase Ib/II study. The purpose of phase Ib is to evaluated the safety, tolerability, pharmacokinetics, immunogenicity, and preliminary antitumor activity of SHR-A1811 in combination with chemotherapy and/or immunotherapy in HER2 expression advanced/metastatic gastric/gastroesophageal junction adenocarcinoma patients.

The Phase II study was designed to evaluate the efficacy and safety of SHR-A1811 in combination with chemotherapy and/or immunotherapy for advanced/metastatic HER2 expression gastric/gastroesophageal conjunctional adenocarcinoma patients.

ELIGIBILITY:
Inclusion Criteria:

1. Age from 18 to 75, Male and female participants
2. Local advanced unresectable or metastatic disease Pathologically documented adenocarcinoma of gastric or gastroesophageal junction;
3. HER2 expression ;
4. Phase Ib: Failed or intolerant to prior standard treatment, or did not receive any systemic anti-tumor therapy; Phase II: previously untreated patients;
5. ECOG 0-1;
6. The expected survival ≥3 months;
7. Sufficient bone marrow and organ functions;

Exclusion Criteria:

1. There were ascites, pleural effusion and pericardial effusion that needed to be treated;
2. Major surgery was performed within 4 weeks;
3. Have active autoimmune disease or history of autoimmune disease;
4. Patients with interstitial pneumonia;
5. There was severe infection within 4 weeks before starting the study treatment;
6. Patients with active pulmonary tuberculosis infection history within 1 year before enrollment;
7. Serious cardiovascular and cerebrovascular diseases;
8. Gastrointestinal perforation and/or gastrointestinal fistula occurred within 6 months before enrollment;

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 258 (Estimated)
Dates: Start 2023-03-14 (Actual); Primary Completion 2027-12 (Estimated); Study Completion 2027-12 (Estimated)

PRIMARY OUTCOMES:
Phase Ib: Dose limiting toxicity (DLT) rates, Occurrence of adverse events (AEs), and serious adverse events (SAEs) | Safety will be assessed for approximately 24 months from informed consent
Phase II: Objective Response Rate (ORR)[ | An average of approximately 12 months

SECONDARY OUTCOMES:
ORR（Phase Ib） | An average of approximately 12 months
DoR（Phase Ib） | An average of approximately 18 months
PFS（Phase Ib） | An average of approximately 18 months
OS（Phase Ib） | An average of approximately 30 months
DoR（Phase II） | An average of approximately 18 months
PFS（Phase II） | An average of approximately 18 months
OS（Phase II） | An average of approximately 30 months
Occurrence of adverse events (AEs), and serious adverse events (SAEs) （Phase II） | Safety will be assessed for approximately 24 months from informed consent]

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Hospital, FuDan University, Shanghai, Shanghai Municipality, China

IPD SHARING:
Plan to Share IPD: Undecided